CLINICAL TRIAL: NCT03924050
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Study of Pemetrexed + Platinum Chemotherapy With or Without Toripalimab (JS001) in Advanced Non-small Cell Lung Cancer (NSCLC) Participants With TKI-resistant EGFR-mutated Tumors
Brief Title: Toripalimab Plus Pemetrexed+Platinus in Advanced Non-small-cell Lungcancer Patients Previsouly Treated EGFR-TKI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-CT25-III-NSCLC
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TORIPALIMAB combined with standard chemotherapy (Experimental)
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 )
- Group Placebo combined with standard chemotherapy (Placebo Comparator)
  Interventions: Drug: TORIPALIMAB INJECTION(JS001 )

INTERVENTIONS:
Drug: TORIPALIMAB INJECTION(JS001 ) — TORIPALIMAB INJECTION(JS001 ) or Placebo, 240mg/6ml/vial, Q3W,up to 2 years of treatment.

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Study to evaluate the efficacy and safety of Toripalimab injection (JS001) or placebo combined with chemotherapy in Advanced Non-small Cell Lung Cancer (NSCLC) Participants with TKI-resistant EGFR-mutated Tumors; and evaluate the population with the best predictive biomarkers, i.e., positive diagnosis population.

About 440 subjects with advanced non-small cell lung cancer with activated EGFR mutation will be 1:1 randomized into two groups, JS001 combined with the standard 1st-line chemotherapy will be given in the study group whereas placebo combined with standard 1st-line chemotherapy will be given in the control group. The stratification will be based on the following factors:

The history of the previous lines of EGFR-TKI treament ( 1st or 2nd generation of TKI vs. 3rd generation of TKI vs. 1st or 2nd generation of TKI + 3rd generation of TKI) ; Disease stage (IIIB-C vs. IV);

ELIGIBILITY:
Inclusion Criteria:

Only the patients meeting all the following criteria can be eligible to participate in the trial:

* Fully informed consent and signed ICF;
* Age of 18-75 years;
* Histologically and/or cytologically confirmed advanced or recurrent stage III B-C or IV (AJCC Version 8) NSCLC with TKI-resistant EGFR-mutated tumors, which also satisfy following conditions: Without T790M mutation in exon 20 after 1st or 2nd generation EGFR-TKI (eg, gefitinib, erlotinib, icotinib, afatinib,etc.) treatment failure;If with T790M mutation in exon 20 after 1st or 2nd generation EGFR-TKI (eg, gefitinib, erlotinib, icotinib, afatinib,etc.),participants are required to have osimertinib or other 3rd generation EGFR-TKI treatment failure prior to enrollment.Participants with osimertinib treatment failure as 1st line therapy (regardless of their EGFR T790M mutation status);Previous neoadjuvant/adjuvant chemotherapy is allowed, but the time interval between the last dose of chemotherapy and recurrence/metastasis must be at least 6 months.
* With at least one measurable disease per RECIST 1.1;
* Agree to provide formalin fixed tumor specimen after EGFR-TKI treatment failure or provide fresh biopsy tissue;
* ECOG performance status of 0-1;
* Life expectancy ≥ 3 months;
* Good organ function;
* Any adverse event resulting from prior treatment, surgery, or radiotherapy must return to grade 0 or 1 according to NCI-CTCAE v5.0, except for alopecia of any grade;
* Willing and able to follow protocol visits, treatment plans, laboratory tests and other study procedures;
* Women of childbearing potential must have negative serum pregnancy test within 3 days prior to the first dose of investigational product:

Exclusion Criteria:

* Exclusion of tumor histology or cytology confirmed the presence of small cell lung cancer components, or squamous cell carcinoma components of more than 10%;
* Combined with other driver mutations with known therapeutic drug, including but not limited to: ALK rearrangement, ROS1 mutation, BRAF600E mutation;
* Previous systematic chemotherapy for advanced NSCLC;
* Subjects with no measurable lesions;
* Subjects with cancer meningitis and spinal cord compression;
* Subjects with untreated central nervous system (CNS) tumor metastasis;
* Subjects were previously treated with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 agent;
* Subjects with any active, known or suspected autoimmune disease;
* Subjects who are now participating in other clinical studies or the last dose of prior investigational drug was given in < 4 weeks (or 5 half-lives) from the first investigational product administration of this study;
* Subjects who were expected to receive any other antitumor therapy (eg, other maintenance therapy for NSCLC, radiotherapy, and/or surgical excision);
* Subjects who received major surgery within 4 weeks prior to enrollment or were not fully recovered from prior surgery;
* Subjects with other malignancies requiring concurrent treatment;
* Subjects with grade II or above myocardial ischemia or myocardial infarction, or subjects with arrhythmia with poor control;
* Subjects with uncontrolled pleural/pericardial effusion, or with ascites requiring repeated drainage;
* Subjects with uncontrolled tumor-related pain;
* Subjects with severe allergic reactions to other monoclonal antibodies and subjects with severe allergic reactions to pemetrexed, platinum or its prophylaxis;
* Subjects with psychological disorder, alcohol alcoholism, drug abuse or drug dependency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-07-17 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
OS | Approximately 5 years
  Overall survival，It's suitable for all subjects.

SECONDARY OUTCOMES:
PFS (Progression Free Survival) by investigator | Approximately 4 years
  Progression free survival (PFS) evaluated by investigators according to the response evaluation criteria in solid tumors (RECIST 1.1)
ORR (Objective Response Rate) | Approximately 4 years
  Objective response rate (ORR) evaluated by investigators based on RECIST1.1;
DOR (Duration of Response) | Approximately 4 years
  Duration of response (DOR) evaluated by investigators and BIRC based on RECIST1.1;
DCR (Disease of Response) | Approximately 4 years
  Disease control rate (DCR) evaluated by investigators based on RECIST1.1;
TTR (Time to Response) | Approximately 4 years
  Time to response (TTR) evaluated by investigators based on RECIST1.1;
Incidence of AEs/SAEs | Approximately 5 years
  Adverse events (AEs) study drug related; serious adverse events (SAEs)study drug related; abnormal value of Lab test according to NCI-CTCAE V5.0

OTHER OUTCOMES:
pd-l1 mutation rate | Approximately 4 years
  To explore the correlation between pd-l1 mutation and efficacy in subjects
immune cell classification | Approximately 5 years
  To explore the correlation between immune cell classification and therapeutic effect

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Peking University Shenzhen Hospital, Shenzhen

REFERENCES:
- [Derived] Jiang T, Wang P, Zhang J, Zhao Y, Zhou J, Fan Y, Shu Y, Liu X, Zhang H, He J, Gao G, Mu X, Bao Z, Xu Y, Guo R, Wang H, Deng L, Ma N, Zhang Y, Feng H, Yao S, Wu J, Chen L, Zhou C, Ren S. Toripalimab plus chemotherapy as second-line treatment in previously EGFR-TKI treated patients with EGFR-mutant-advanced NSCLC: a multicenter phase-II trial. Signal Transduct Target Ther. 2021 Oct 15;6(1):355. doi: 10.1038/s41392-021-00751-9. PMID 34650034